CLINICAL TRIAL: NCT03057184
Title: Behavioral Intervention to Reduce Resistance in Those Attending Adult Day Care Centers: PROCENDIAS Study. A Randomized Clinical Trial
Brief Title: Behavioral Problems Related to Attendance Adult Day Care Centers
Acronym: PROCENDIAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Collaborators: Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GRS1274/B/16
Record Dates: First submitted 2017-02-12; First posted 2017-02-17 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Family Members; Dependence
Keywords: Adult Day Care Center; behavioral problems; caregivers
MeSH Terms: conditions — Problem Behavior | interventions — Methods

STUDY DESIGN:
Intervention Model Description: It is an experimental design using random assignment to select 130 family members responsible for the preparation and transfer of the care-recipient from their home to the ADCC: was randomized to an intervention group or control group (care as usual).
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): behavioral intervention program
  Interventions: Behavioral: Intervention
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Intervention — The intervention will consist of 8 weekly sessions, with a duration of 90 minutes. Although each intervention is adapted to the specific behavioral problems
  Arms: Intervention group

SUMMARY:
Adult Day Care Centers (ADCC) offer important relief and rest services for family caregivers. However, some caregivers report that behavioral and psychological symptoms of dementia (BPSD) arise when they prepare dependents for the ADCC, especially when they have dementia. This issue increases stress for caregivers and contributes to a worsening of their mental health and quality of life. The present study evaluates the effectiveness of a behavioral intervention program aimed at reducing the reluctance of the dependent to attend the ADCC. We hope that reducing resistance will have a positive influence on the mental health of caregivers.

DETAILED DESCRIPTION:
Randomized controlled trial. The protocol was performed in accordance with the SPIRIT 2013 Statement and was registered in the Clinical Trials-gov (PROCENDIAS study). The CONSORT guidelines were rigorously followed in this randomized clinical trial. Information about the study, including the objectives, procedures, possible benefits and risks was provided at the beginning of the study and written informed consent, according to the general recommendations of the Declaration of Helsinki (World Medical, 2013), was obtained from each study participant.

Study Population:

The study was conducted in the municipality of Salamanca based on a list of people who attend an ADCC and whose relatives agree to participate voluntarily in the study. The reference population will be people attending ADCC and the relatives who participate in their care and who identify themselves as principal caregivers for this task.

Variables and measurement instruments The data will be collected in an interview, using the questionnaire designed for the study.

1. Outcome variables:

   Caregiviers:

   Sociodemographic information. The frequency and distress associated with disruptive behaviors was measured with the Spanish version of the disruptive behaviors sub-scale of the Revised Memory and Behavior Problems Checklist (RMBPC), an 8-item scale with answers ranging from 0 (never occurred) to 4 (occurs daily or more often), for the frequency score, and from 0 (not at all) to 4 (extremely), for the distress score.

   Caregivers' mental health as self-perceived by caregivers was measured using the 12-item version of the GHQ-12 (Goldberg & Hillier, 1979). Depressive symptomatology was measured through the Center for Epidemiologic Studies Depression Scale (CES-D; Radloff, 1977), a 20-item scale. Caregiver stress and overload were measured through the short Zarit Burden Interview (short ZBI; Gort et al., 2005). Family function has been measured using the family APGAR test (Smilkstein, 1978).
2. ADCC Users:

Sociodemographic variables: age, gender, marital status and years of schooling; comorbidity (Charlson's comorbidity index). Functional capacity: basic activities of daily life (Barthel index); instrumental activities of daily living (Lawton-Brody index);

Baseline Evaluation and Follow-Up:

All ADCCs in the city were invited to participate in the study and those centres agreeing to do so sent an information letter about the project to the home of each of their users inviting them to participate in the study. Caregivers who agreed to participate reported at their centre and the centre contacted the research team. Participants received a telephone call from the research team after about 10-15 days to arrange an appointment and perform the baseline evaluation. The assessments were made either at the ADCC or at the relevant health centre. Those that met the inclusion criteria were subsequently selected. Once this phase was finished, the caregiver was assigned to the intervention group (IG) or control group (CG), in accordance with a previously randomised sequence. The assignment sequence was generated by an independent researcher using Epidat 4.2 software (Consellería de Sanidade, 2016) with a 1:2 a ratio. The selected family caregivers were informed that a weekly session of 90 minutes would be held over a period of 8 weeks in groups of 8-10 participants each. Caregivers of relatives with different pathologies were included. The same evaluation was performed for the CG and the IG at baseline and at 6 months after randomisation.

ELIGIBILITY:
Inclusion Criteria:

1. Participants in the study are those family members who help in the care of the person attending the ADCC at least two days a week;
2. Family caregivers perform or participate in organizing the dependent patient's preparation to visit the ADCC, with or without the help of another person. It is define "preparation for attendance" as all the activities performed by the caregivers in interaction with the patient, from the moment in which they begin to prepare until they get into the vehicle taking them to the ADCC, with the aim of facilitating their ADCC attendance. This includes, for example, waking them up, getting them out of bed, helping them shower and get dressed, assisting them at breakfast, helping them to walk and use the stairs, communicating with them about current actions and what they will be doing in the immediate future;
3. Family caregivers recognize the existence of at least one BPSD associated with ADCC care;
4. Signature of informed consent by family caregivers.

Exclusion Criteria:

1. Paid caregivers;
2. Family caregivers who do not participate in the preparation for the ADCC visit;
3. Those who do not sign informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-02-12 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
disruptive behaviors | Post intervention (6 months follow-up assessment will be performed)
  Measured by the questionary disruptive behaviors will be measured with RMBPC

CONTACTS AND LOCATIONS:
Overall Officials: Luis Garcia Ortiz, MD, Study Director — Instituto de Investigación Biomédica de Salamanca
Locations (1):
- Fundacion INFOSALUD, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided